CLINICAL TRIAL: NCT01998386
Title: Tooth Whitening With Hydrogenperoxide in Adolescents - Controlled Clinical Trial
Brief Title: Tooth Whitening With Hydrogenperoxide in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TWHPA
Record Dates: First submitted 2013-09-15; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Posteruptive Color Change of Tooth
Keywords: Tooth Whitening; Adolescent; Clinical Trial
MeSH Terms: interventions — Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo gel without hydrogen peroxide (Placebo Comparator): The volunteers of this group will receive a placebo gel without hydrogen peroxide for whitening treatment.
  Interventions: Other: Placebo gel without hydrogen peroxide
- 6.0% hydrogen peroxide - White Class (Experimental): Volunteers of this group will receive a gel with 6.0% hydrogen peroxide - White Class with calcium for whitening treatment.
  Interventions: Other: 6.0% hydrogen peroxide - White Class
- 7.5% hydrogen peroxide - White Class (Experimental): The volunteers of this group will receive a gel with 7.5% hydrogen peroxide -White Class with calcium for whitening treatment.
  Interventions: Other: 7.5% hydrogen peroxide - White Class
- 7.5% hydrogen peroxide - Oral-B 3D White (Experimental): The participants in this group will receive disposable whitening strips - Oral-B 3D White for whitening treatment.
  Interventions: Other: 7.5% hydrogen peroxide - Oral-B 3D White

INTERVENTIONS:
Other: Placebo gel without hydrogen peroxide — Castings will be made of the upper and lower arches of the volunteers and plaster will be poured into the molds. Individual plastic molds (vacuum form, flexible acetate 1 mm in thickness) will be made for each arch using the plaster models. After fitting the molds in the oral cavity, the volunteers will receive oral and written instructions on how to use the whitening gel and will be instructed to perform proper oral hygiene with dental floss and a tooth brush prior to the application of the whitening agent. The volunteers will be instructed to use the molds with the gel one hour a day for seven days. Thirty days after the beginning of treatment, the volunteers in this group will receive the whitening treatment with 6.0% hydrogen peroxide - White Class with calcium.
  Arms: Placebo gel without hydrogen peroxide
Other: 6.0% hydrogen peroxide - White Class — Castings will be made of the upper and lower arches of the volunteers and plaster will be poured into the molds. Individual plastic molds (vacuum form, flexible acetate 1 mm in thickness) will be made for each arch using the plaster models. After fitting the molds in the oral cavity, the volunteers will receive oral and written instructions on how to use the whitening gel 6.0% hydrogen peroxide - White Class with calcium and will be instructed to perform proper oral hygiene with dental floss and a tooth brush prior to the application of the whitening agent. The volunteers will be instructed to use the molds with whitening gel one hour a day for seven days.
  Arms: 6.0% hydrogen peroxide - White Class
Other: 7.5% hydrogen peroxide - White Class — Castings will be made of the upper and lower arches of the volunteers and plaster will be poured into the molds. Individual plastic molds (vacuum form, flexible acetate 1 mm in thickness) will be made for each arch using the plaster models. After fitting the molds in the oral cavity, the volunteers will receive oral and written instructions on how to use the whitening gel 7.5% hydrogen peroxide - White Class with calciumand will be instructed to perform proper oral hygiene with dental floss and a tooth brush prior to the application of the whitening agent. The volunteers will be instructed to use the molds with whitening gel one hour a day for seven days.
  Arms: 7.5% hydrogen peroxide - White Class
Other: 7.5% hydrogen peroxide - Oral-B 3D White — The participants in this group will receive four disposable whitening 7.5% hydrogen peroxide - Oral-B 3D White strips for daily individual use. The volunteers will be instructed to perform proper oral hygiene with dental floss and a tooth brush prior to the application of the whitening strips. The volunteers will receive oral and written instructions on how to use the whitening strips, which will be placed on the surface of the teeth for 30 minutes twice a day for seven days.
  Arms: 7.5% hydrogen peroxide - Oral-B 3D White

SUMMARY:
The specific objective of this study is:

* Evaluate and quantify colorimetric changes in young permanent anterior teeth;
* Compare the efficiency and efficacy of three gels used for self-administered home whitening and an over the counter whitening strip;
* Analyze the increase in dental sensitivity in adolescent patients submitted to home whitening with 6% and 7.5% hydrogen peroxide with and without the addition of calcium (whitening strips);
* Assess sensitivity, comfort and acceptance of whitening strips by patients;
* Assess patient satisfaction with the method and material used for home whitening.

DETAILED DESCRIPTION:
The aim of the proposed controlled clinical trial will be to assess colorimetric changes and increased dental sensitivity in adolescent patients submitted to tooth whitening with 6% and 7.5% hydrogen peroxide using home kits with whitening strips. Adolescents aged 12 to 20 years will be allocated to different groups based on treatment (n = 16 per group): 1) placebo; 2) 6.0% hydrogen peroxide (White Class with calcium - FGM); 3) 7.5% hydrogen peroxide (White Class with calcium - FGM); and 4) 7.5% hydrogen peroxide (Oral B 3D White - Oral-B). After the whitening procedures, the participants will be evaluated using a visual analogue scale for tooth sensitivity and digital spectrophotometry for the measurement of changes in color.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 20 years; diagnosis of altered color on maxillary and mandibular anterior teeth with initial color equivalent to A2 on the Vita scale (Vita Zahnfabrik); signed statement of informed consent

Exclusion Criteria:

* Dental anomalies (malformation, carious lesions, fractures); presence of at least four maxillary and/or mandibular anterior teeth; known adverse reaction to peroxide; use of whitening agents (administered in dental office or at home) in the previous year; currently undergoing orthodontic treatment, orthopedic treatment of the jaws or psychological treatment; use of medication that can alter the color of the teeth, such as ferrous sulfate.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Discoloration | Change of teeth color after 7 days of the beginning of treatment
  Color readings of the vestibular region of the maxillary and mandibular anterior teeth will be performed by a previously trained examiner blinded to the allocation of the volunteers to the different groups. A digital spectrophotometer will be used for the colorimetric evaluation.
  It will be carried out in all groups at the following times: pre-treatment period, immediately following the first treatment period, after seven days, after 30 days, after six months, after 12 months, after 24 months, and after 48 months.

SECONDARY OUTCOMES:
Dental sensitivity | Sensivity alteration after 7 days of the beginning of treatment
  The volunteers will inform the degree of sensitivity at all evaluation times using a visual analog scale ranging from 0 (absence of sensitivity) to 10 (maximum sensitivity).
  Evaluations of dental sensitivity will be carried out in all groups at the following times: pre-treatment period, immediately following the first treatment period, after seven days, after 30 days, after six months, after 12 months, after 24 months and after 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Bussadori, Principal Investigator — University of Nove de Julho; Marcelo M Pinto, Study Chair — University of Nove de Julho; Camila HL Godoy, Study Chair — University of Nove de Julho; Rubia G Lopes, Study Chair — University of Nove de Julho; Zenildo S Silva Junior, Study Chair — University of Nove de Julho; Silvia RG Olivan, Study Chair — University of Nove de Julho; Lara J Motta, Study Chair — University of Nove de Julho; Olga M Altavista, Study Chair — University of Nove de Julho; Katia Lumi, Study Chair — University of Nove de Julho; Ana Paula T Sobral, Study Chair — FGM
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Pinto MM, Goncalves ML, Mota AC, Deana AM, Olivan SR, Bortoletto C, Godoy CH, Vergilio KL, Altavista OM, Motta LJ, Bussadori SK. Controlled clinical trial addressing teeth whitening with hydrogen peroxide in adolescents: a 12-month follow-up. Clinics (Sao Paulo). 2017 Mar;72(3):161-170. doi: 10.6061/clinics/2017(03)06. PMID 28355362
- [Derived] Pinto MM, de Godoy CH, Bortoletto CC, Olivan SR, Motta LJ, Altavista OM, Lumi K, Sobral AP, Bussadori SK. Tooth whitening with hydrogen peroxide in adolescents: study protocol for a randomized controlled trial. Trials. 2014 Oct 14;15:395. doi: 10.1186/1745-6215-15-395. PMID 25315893